CLINICAL TRIAL: NCT04358861
Title: Healing Outcome of Nonsurgical Root Canal Treatment in Maxillary Molars With Dental Operating Microscope : A Randomized Controlled Trial
Brief Title: Healing Outcome of Root Canal Therapy in Maxillary Molars With DOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Neelam
Record Dates: First submitted 2020-04-17; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Periapical Periodontitis
Keywords: Dental Operating Microscope
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Nonsurgical Root canal therapy was performed using dental operating microscope in the experimental group.
  Interventions: Procedure: Nonsurgical Root canal therapy; Device: Dental operating microscope
- Control group (Active Comparator): Nonsurgical Root canal therapy was performed without any magnification aid in control group.
  Interventions: Procedure: Nonsurgical Root canal therapy

INTERVENTIONS:
Procedure: Nonsurgical Root canal therapy — After administration of LA and rubber dam isolation, acess cavity was prepared using carbide burs. Working length was determined using root ZX apex locator and was verified radiographically. Canal preparation was done with protaper gold rotary instruments. 5ml of 5.25% NaOCl was used as irrigant. After instrumentation , the canals were irrigated with 5.0 ml of 17% EDTA for 1minute followed by irrigation with 5.0 ml of 5.25% NaOCl. Canals were dried with absorbent paper points, filled with calcium hydroxide paste and access cavity was restored with IRM.At the recall appointment ; after one week,paste removal, copious irrigation was done with 5.25% NaOCl and canals were dried with paper points. Canals were obturated with Gutta-Percha and ZOE based sealer.
Device: Dental operating microscope — Dental operating microscope; a high magnification and illumination device was used in experimental group for performing nonsurgical root canal therapy.
  Arms: Experimental group

SUMMARY:
The aim of study was to evaluate the effect of dental operating microscope use on the healing outcome of non surgical endodontic treatment of maxillary molars.

DETAILED DESCRIPTION:
Prior to treatment a thorough clinical and radiological examination was carried out. A thorough history was taken from each patient and written informed consent was taken after explaining the procedure, risks and benefits. Mature maxillary first permanent molar with diagnosis of periapical periodontitis (as confirmed clinically & by periapical radiograph) was chosen for the study. Fifty participants were randomly assigned to either the dental operating microscope group or to control group (without using dental operating microscope) for the treatment.

After administration of local anesthesia and rubber dam isolation of the involved tooth ; access cavity was prepared using carbide bur and refined using ultrasonic tip in both groups. In both the groups similar protocol for irrigation, obturation and post operative restorations was followed. Immediate post-operative radiograph was taken using preset exposure parameters and follow up clinical and radiographic examination was carried at 12th month.

ELIGIBILITY:
Inclusion Criteria:

* Patient willing to participate in the study
* Age > 18 years
* Maxillary permanent first molar having apical periodontitis requiring primary endodontic treatment
* Radiographic evidence of periapical radiolucency (minimum size 2 mmx 2 mm) and a diagnosis of pulpal necrosis as confirmed by negative response to cold and electrical tests and absence of bleeding on entering the pulp chamber

Exclusion Criteria:

* Unwillingness of patient.
* Retreatment cases
* Presence of internal or external resorption ,root canal perforations during endodontic treatment and immature teeth.
* Periodontally compromised teeth
* Immunocompromised, diabetic, pregnant and hypertensive patients
* Vertical root fractures
* Teeth those are not suitable for rubber dam application

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Clinical and radiographic success | 12 months
  long term clinical and radiographic success measured in terms of reduction in size of periapical radiolucency on radiograph from baseline to 12 months using PAI score 1,2 as healing and more than 2 as non healing

SECONDARY OUTCOMES:
Number of canals located in MB root | 12 months
  incidence of additional canals located in MB root

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: Undecided